CLINICAL TRIAL: NCT06488079
Title: Effectiveness of Front-of-Pack Nutritional Labels in Promoting Greater Adherence to the Mediterranean Diet
Brief Title: Effectiveness of Different Front-of-Pack Nutritional Labels in Promoting Greater Adherence to the Mediterranean Diet Among Italian Consumers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donini Lorenzo M (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor-Investigator, Donini Lorenzo M, Full Professor, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CERT_18F2F1CDB00
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutri-Score label (Experimental)
  Interventions: Other: Summary Label
- NutrInform Battery label (Experimental)
  Interventions: Other: Nutrient-specific label
- No label (Sham Comparator)
  Interventions: Other: No label

INTERVENTIONS:
Other: Summary Label — The Nutri-Score Front-of-Pack nutritional label
  Arms: Nutri-Score label
Other: Nutrient-specific label — The NutrInform Battery Front-of-Pack nutritional label
  Arms: NutrInform Battery label
Other: No label — Conventional food educational flyer
  Arms: No label

SUMMARY:
The goal of this clinical trial is to learn if Front-of-Pack labels, namely Nutri-Score and NutrInform Battery, work to improve adherence to the Mediterranean diet among healthy Italian adult participants. It will also learn about the label's ability to increase nutritional knowledge and participant's response in terms of orthorexic behaviour. The main questions it aims to answer are:

* Does FOP nutritional labels work to guide participants' food choices towards healthier diets?
* Do they increase participants' nutritional knowledge?
* To what extent are they related to obsessive focus on healthy eating, such as orthorexia nervosa? Researchers will compare the labels to a no label condition (in which participants were only given a conventional nutrition education flyer) to see if labels work to improve healthiness in individual diets.

Participants will:

* Complete an initial questionnaire's battery
* Use the assigned FOP label every day for 1 month to orient their food choices
* Answer to final questionnaires

ELIGIBILITY:
Inclusion Criteria:

* limited to participants older than 18 years

Exclusion Criteria:

* people currently on a diet for religious/ethical/personal choice or medical prescription
* people with a degree or a professional expertise in the area of field, nutrition, and physical exercise
* people who know one of the interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3029 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet | 30 days
  The adherence is measured with the PREDIMED (PREvención con DIeta MEDiterránea) PLUS questionnaire adapted for the Italian population. The questionnaire asks about the frequency of consumption of traditional Mediterranean food (daily or weekly) by defining the portion size, or asking about the use of food with "yes or no" options, or identifying preferences between different food options. Possible values range from 0 to 17. Higher values correspond to a higher adherence.

SECONDARY OUTCOMES:
Nutrition Knowledge | 30 days
  Nutrition knowledge is measured by the General Nutrition Knowledge Questionnaire (GNKQ) adapted for the Italian population (I-NK Questionnaire). It is composed of four sections exploring different aspects of NK: (NK1) Experts' recommendations (9 questions); (NK2) Food composition (10 questions); (NK3) Food choices and nutrition labels (11 questions); (NK4) Diet-disease associations (16 questions). Possible values range from 0 to 88. Higher values correspond to a higher knowledge.
Orthorexic behaviour | 30 days
  Orthorexic behaviour is measured by the ORTO-R Questionnaire. The ORTO-R is an adaptation of the ORTO-15, from which it contains six items which were identified as the best markers of orthorexia nervosa. The response scale is a five-point Likert-type scale and a higher score reflects higher intensity of orthorexia nervosa thoughts and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Maria Donini, Principal Investigator — Sapienza University
Locations (1):
- Sapienza University, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
By decision of the ethics committee data can be shared only in an aggregated form